CLINICAL TRIAL: NCT02819531
Title: A Single Center, Randomized Trial of Treatment Strategies for Obstructive Calcified Coronary Lesions: Efficacy CompariSon of Pre-stenting Atherectomy Versus Scoring ballooN for calcifieD Coronary Lesions Coronary Lesions (ECSPAND)
Brief Title: Efficacy CompariSon of Pre-stenting Atherectomy Versus Scoring ballooN for calcifieD Coronary Lesions Coronary Lesions
Acronym: ECSPAND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Emmanouil Brilakis, Director of Cardiac Catheterization Laboratories, Professor of Medicine, North Texas Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-017
Record Dates: First submitted 2016-06-21; First posted 2016-06-30 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Atherosclerosis; Coronary Artery Disease
Keywords: Coronary Atherectomy; percutaneous coronary intervention
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease | interventions — Atherectomy, Coronary

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rotational atherectomy (Active Comparator): RA protocol: After IVUS protocol, patients who are randomized to RA will undergo coronary wiring of the target lesion and subsequent advancement of the RA burr. The RA system is performed using standard technique under intravenous infusion of heparin. The atherectomy burr size will be determined by the operator.
  Interventions: Device: Rotational atherectomy
- Orbital atherectomy (Active Comparator): OAS protocol: After IVUS protocol, patients who are randomized to OAS will undergo coronary wiring of the target lesion and subsequent advancement of the OAS according to the manufacturer's guidelines.
  Interventions: Device: Orbital atherectomy
- Scoring balloon system (Active Comparator): SBS protocol: After IVUS protocol, patients who are randomized to SBS will undergo coronary wiring of the target lesion and balloon inflation with SBS performed by standard technique under intravenous infusion of heparin. SBS will be used according to the manufacturer's guidelines.
  Interventions: Device: Scoring balloon system

INTERVENTIONS:
Device: Rotational atherectomy — Pre-stenting lesion modification using the rotational atherectomy device using standard technique under intravenous infusion of heparin. Burr size will be selected by the operator according to vessel size. IVUS images will be obtained before lesion modification and after stenting.
  Arms: Rotational atherectomy
Device: Orbital atherectomy — Pre-stenting lesion modification using the orbital atherectomy device according the manufacturer's guidelines. IVUS images will be obtained before lesion modification and after stenting.
  Arms: Orbital atherectomy
Device: Scoring balloon system — Pre-stenting lesion modification using the scoring balloon system according the manufacturer's guidelines. IVUS images will be obtained before lesion modification and after stenting.
  Arms: Scoring balloon system

SUMMARY:
Design: The proposed study is a randomized study comparing the relative effectiveness of three lesion modification strategies (RA, SBS, or OAS) in the treatment of obstructive CCLs using the change in lumen size measurements (MLA, RLA, MSA and the ratio of MSA/MLA) obtained with IVUS or OCT. Patients will be blinded to treatment assignment for the duration of the study.

Treatment: Patients who are randomized to RA will undergo coronary wiring of the CCL and subsequent advancement of the RA burr. The RA system is performed using standard technique under intravenous infusion of heparin. The atherectomy burr size will be determined by the operator.

Patients who are randomized to OAS will undergo coronary wiring of the CCL and subsequent advancement of the OAS according to the manufacturer's guidelines.

Control: Patients who are randomized to SBS will undergo coronary wiring and balloon inflation with SBS performed by standard technique under intravenous infusion of heparin. SBS will be used according to the AngioSculpt manufacturer's guidelines.

Duration: 30 days follow-up.

The primary trial objective is to determine which of the three treatment strategies for treating calcified coronary lesions (RA, SBS, or OA) is superior for obtaining higher ratio of final in-stent minimum lumen area/reference lumen area, as determined by IVUS or OCT (primary study endpoint).

The secondary objectives are to compare the following:

1. Difference in pre- vs. post-treatment minimum lumen area (MLA, lumen area gain), as determined by IVUS or OCT (secondary endpoint)
2. Mean final minimal stent area (MSA), as assessed by IVUS or OCT (secondary endpoint)
3. Ratio of final in-stent minimum lumen diameter/reference lumen diameter, as determined by quantitative coronary angiography (secondary endpoint)
4. Incidence of major adverse cardiac events (death, myocardial infarction, target vessel revascularization) during 30 days of follow-up (secondary endpoints)
5. Procedure time, fluoroscopy time, and contrast volume (secondary endpoints)

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Clinical indication for coronary intervention such as ischemic symptoms and/or a positive functional study
3. Found to have a de novo severe calcification (radio opacities noted without cardiac motion on contrast injection, lesion length >15 mm, or presence of >270° calcification on one cross-sectional view of IVUS) in a native coronary artery on fluoroscopy or IVUS

Exclusion Criteria:

1. Subject is currently participating in an investigational device or pharmaceutical treatment protocol
2. Persistent (>10 minutes) hypotension (systolic blood pressure <90 mmHg)
3. Need for revascularization of multiple lesions during the index PCI
4. Unprotected left main (>50%) or equivalent left main disease
5. Non-calcified lesions
6. Chronic total occlusions, extreme lesion tortuosity including Type B/C lesions
7. Severe left ventricular dysfunction (ejection fraction <25%)
8. History of bleeding diathesis or coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Ratio of final in-stent minimum lumen area/reference lumen area | Immediately after stenting
  IVUS measurement based determination of ratio of final in-stent minimum lumen area/reference lumen area, as determined by IVUS

SECONDARY OUTCOMES:
Difference in pre- vs. post-treatment minimum lumen area (MLA, lumen area gain) | Immediately after stenting
  IVUS measurement based determination of difference in pre- vs. post-treatment minimum lumen area (MLA, lumen area gain)
Mean final minimal stent area (MSA) | Immediately after stenting
  IVUS measurement based determination of Mean final minimal stent area (MSA)
Ratio of final in-stent minimum lumen diameter/reference lumen diameter | Immediately after stenting
  Quantitative coronary angiography based determination of ratio of final in-stent minimum lumen diameter/reference lumen diameter
Lower incidence of major adverse cardiac events (death, myocardial infarction, target vessel revascularization) during 30 days of follow-up | 30 days
Procedure time | Immediately after the end of the interventional procedure
Fluoroscopy time | Immediately after the end of the interventional procedure
Contrast volume | Immediately after the end of the interventional procedure

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil S Brilakis, MD, PhD, Study Chair — North Texas Veterans Healthcare System; Jerrold Grodin, MD, Principal Investigator — North Texas Veterans Healthcare System

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Genereux P, Lee AC, Kim CY, Lee M, Shlofmitz R, Moses JW, Stone GW, Chambers JW. Orbital Atherectomy for Treating De Novo Severely Calcified Coronary Narrowing (1-Year Results from the Pivotal ORBIT II Trial). Am J Cardiol. 2015 Jun 15;115(12):1685-90. doi: 10.1016/j.amjcard.2015.03.009. Epub 2015 Mar 24. PMID 25910525
- [Background] Vaquerizo B, Serra A, Miranda F, Triano JL, Sierra G, Delgado G, Puentes A, Mojal S, Brugera J. Aggressive plaque modification with rotational atherectomy and/or cutting balloon before drug-eluting stent implantation for the treatment of calcified coronary lesions. J Interv Cardiol. 2010 Jun;23(3):240-8. doi: 10.1111/j.1540-8183.2010.00547.x. PMID 20636844
- [Background] Adamian M, Colombo A, Briguori C, Nishida T, Marsico F, Di Mario C, Albiero R, Moussa I, Moses JW. Cutting balloon angioplasty for the treatment of in-stent restenosis: a matched comparison with rotational atherectomy, additional stent implantation and balloon angioplasty. J Am Coll Cardiol. 2001 Sep;38(3):672-9. doi: 10.1016/s0735-1097(01)01458-9. PMID 11527615
- [Background] Genereux P, Madhavan MV, Mintz GS, Maehara A, Palmerini T, Lasalle L, Xu K, McAndrew T, Kirtane A, Lansky AJ, Brener SJ, Mehran R, Stone GW. Ischemic outcomes after coronary intervention of calcified vessels in acute coronary syndromes. Pooled analysis from the HORIZONS-AMI (Harmonizing Outcomes With Revascularization and Stents in Acute Myocardial Infarction) and ACUITY (Acute Catheterization and Urgent Intervention Triage Strategy) TRIALS. J Am Coll Cardiol. 2014 May 13;63(18):1845-54. doi: 10.1016/j.jacc.2014.01.034. Epub 2014 Feb 19. PMID 24561145